CLINICAL TRIAL: NCT06007950
Title: Impacts of Time-Restricted Eating on Weight, Cardiometabolic and Cardiovascular Health in Patients With Acute Coronary Syndrome
Brief Title: Time-restricted Eating Study (TRES): Impacts on Anthropometric, Cardiometabolic and Cardiovascular Health
Acronym: TRES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Ministry of Higher Education, Malaysia (Other)
Responsible Party: Principal Investigator, MAZUIN KAMARUL ZAMAN, Principal Investigator, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TRES2301
Record Dates: First submitted 2023-08-11; First posted 2023-08-23 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Infarction
Keywords: coronary heart disease; time-restricted eating; intermittent fasting
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Intermittent Fasting

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ad-libitum eating duration (No Intervention): 24 patients will be randomly assigned to the control group. Participants will be asked to continue usual eating duration. Participants will receive the standard care and heart-healthy nutrition education.
- Time-restricted eating (TRE) duration (Experimental): 24 patients will be randomly assigned to the intervention group. Participants in this arm will be asked to limit the number of hours they eat in a day to 10 hours in addition to receiving the standard of care health and heart-healthy nutrition education.
  Interventions: Behavioral: Time-restricted eating 10-hr

INTERVENTIONS:
Behavioral: Time-restricted eating 10-hr — Time-restricted eating is a form of intermittent fasting. In this study, 10-hr TRE will be employed, where eating duration is limited to 10 hours. Participants are allowed to consume non-caloric beverages during fasting period.
  Arms: Time-restricted eating (TRE) duration

SUMMARY:
The goal of this clinical trial is to learn about the effects of time-restricted eating in patients with history of acute coronary syndrome. The main questions it aims to answer are: 1) Is 10-hr TRE safe and feasible for patients with ACS; 2)What are the impacts of 10-hr TRE on anthropometric measurements, cardiometabolic health and cardiovascular health compared to ad libitum eating in patients with ACS?. Participants will be asked to limit eating duration to 10 hours daily.

DETAILED DESCRIPTION:
Justification: The effects of TRE on humans varies results, with some showing improvements in weight loss, insulin sensitivity, and cardiovascular markers, while others exhibiting no significant changes. TRE studies on metabolically altered individuals especially patients with heart diseases are limited.

Written approval of the study has been obtained from the Universiti Teknologi MARA Ethics Committee before commencement of this study.

The TRES study utilizes an investigator-led, pragmatic, parallel, randomized, single-blinded clinical trial design to evaluate the safety, feasibility, and effectiveness of a 10-hour time-restricted eating (TRE) intervention compared to unrestricted eating in patients diagnosed with acute coronary syndrome. The study aims to assess the impact of TRE on anthropometric measurements, as well as cardiometabolic and cardiovascular health outcomes. The duration of the randomized controlled trial (RCT) spans a period of five weeks. The trial consisted of a baseline period of one week, which was then followed by a four-week intervention phase. The participants will be assigned randomly to either the TRE (Time-Restricted Eating) group or the control group, which involves ad libitum eating. They will be instructed to adhere to their allotted eating duration during the four-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18- 65 years old.
* Had history of acute coronary syndrome (ACS)
* Clinically stable
* Self-reported eating window of at least 12 h per day.

Exclusion Criteria:

* Severe obesity (body mass index ≥40 kg m-2).
* Unstable weight in the past three months (gain or lose more than 4 kg of weight).
* Unstable cardiovascular, renal, cardiac, liver, lung, adrenal, or nervous system disease that may compromise study validity.
* Any medications or supplements known to change sleep, circadian rhythms, or metabolism.
* Pregnant or lactating women.
* Perform overnight shift work more than one day/week on average.
* Regularly fasted for more than 15 hours/day or having completed twelve 24-hr fasts within the past three months).
* Active use of tobacco or illicit drug or history of treatment for alcohol abuse.
* Type I diabetes or diabetic, treated with insulin.
* Use of anti-obesity drugs or other drugs affecting body weight.
* Currently enrolled in weight loss or management programme, including surgical intervention.
* Severe kidney failure (glomerular filtration rate (GFR) <30 mL/min).
* Eating disorder or current diagnosis of uncontrolled psychiatric illness, which may impair study involvement.
* Malignancy undergoing active treatment.
* Had gastrointestinal surgery or impaired nutrient absorption.
* Travelled more than two time zones away two months prior to enrolling in the trial or will travel more than two time zones away during the study period.
* Concurrent participation in other interventional studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 4 weeks (pre- & post intervention)
  unit: kg

SECONDARY OUTCOMES:
Change in lean body mass | 4 weeks (pre- & post intervention)
  unit : kg
Change in fat mass | 4 weeks (pre- & post intervention)
  unit : kg
Change in fasting glucose concentration | 4 weeks (pre- & post intervention)
  Glycaemic biomarker, unit: mmol/L
Change in fasting insulin concentration | 4 weeks (pre- & post intervention)
  Glycaemic biomarker, unit:pmol/L
Change in total cholesterol concentration | 4 weeks (pre- & post intervention)
  Lipid metabolism biomarker, unit: mmol/L
Change in high-density lipoprotein concentration | 4 weeks (pre- & post intervention)
  Lipid metabolism biomarker, unit: mmol/L
Change in low-density lipoprotein concentration | 4 weeks (pre- & post intervention)
  Lipid metabolism biomarker, unit: mmol/L
Change in triglycerides concentration | 4 weeks (pre- & post intervention)
  Lipid metabolism biomarker, unit: mmol/L
Change in C-reactive protein concentration | 4 weeks (pre- & post intervention)
  Inflammatory biomarkers, unit: mg/dL
Change in Malondialdehyde (MDA) level | 4 weeks (pre- & post intervention)
  Oxidative stress Lipid peroxidation, unit:μmol/L
Change in flow-mediated dilatation, | 4 weeks (pre- & post intervention)
  Endothelial function, unit:%
Change in Brachial-ankle pulse wave velocity | 4 weeks (pre- & post intervention)
  arterial stiffness, unit:m/s
Change in perceived appetite | 4 weeks (pre- & post intervention)
  Visual analog scale (VAS), linear scale in 100mm (not hungry at all-extremely hungry)
Adverse event monitoring | 4 weeks
  Report of incidence of adverse events for safety monitoring
Change in Hemoglobin level | 4 weeks
  Safety monitoring, unit: g/dl
Change in sleep quality | 4 weeks (pre- & post intervention)
  Pittsburgh Sleep Quality Index (PSQI) scale, A higher score indicates a worse sleep quality. PSQI score >5= poor sleep.
Change in physical activity | 4 weeks (pre- & post intervention)
  Short version of the International Physical Activity Questionnaire (IPAQ), unit: metabolic equivalent (MET)-minutes

OTHER OUTCOMES:
Rate of weekly compliance to intervention | 4 weeks
  Adherence to intervention, number of days complied to eating duration assigned/ 7 daysx100%
Change in caloric intake | 4 weeks (pre- & post intervention)
  Dietary energy consumption, unit: kcal/day

CONTACTS AND LOCATIONS:
Overall Officials: Mazuin Kamarul Zaman, MMed Sc, Principal Investigator — Universiti Teknologi Mara
Locations (1):
- Pusat Perkhidmatan Klinikal (CTC) UiTM, Kuala Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No